CLINICAL TRIAL: NCT06465316
Title: A Phase 1b Trial of Teclistamab in Combination With Iberdomide for Relapsed/Refractory Multiple Myeloma
Brief Title: Testing Teclistamab (TECVAYLI) in Combination With Iberdomide for Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-04754; NCI-2024-04754 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10620 (Other: Dana-Farber - Harvard Cancer Center LAO); 10620 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2024-06-17; First posted 2024-06-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; iberdomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (iberdomide, teclistamab) (Experimental): Patients receive teclistamab SC on days 1, 4, 7, 15 and 22 for cycle 1 and days 1, 8, 15 and 22 for remaining cycles. Patients also receive iberdomide PO QD on days 1-21 for cycle 2 and beyond. Cycles repeat every 28 days for up to 4 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood and urine sample collection, bone marrow aspiration and biopsy and PET/CT or PET/MR throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Iberdomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Teclistamab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Iberdomide — Given PO
  Other Names: CC 220; CC-220
Procedure: Magnetic Resonance Imaging — Undergo PET/MR
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT or PET/MR
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Teclistamab — Given SC
  Other Names: JNJ 64007957; JNJ-64007957; JNJ64007957; Teclistamab-cqyv; Tecvayli

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of iberdomide in combination with teclistamab in treating multiple myeloma that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory). Iberdomide is a medication that belongs to a group of drugs known as cereblon E3 ligase modulators. Iberdomide works by targeting and destroying proteins that help myeloma cancer cells to survive. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as teclistamab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Giving iberdomide in combination with teclistamab may be safe and tolerable in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimate the recommended phase 2 dose (RP2D) of iberdomide in combination with teclistamab.

SECONDARY OBJECTIVES:

I. To evaluate the safety and toxicity profile of iberdomide in combination with teclistamab.

II. To observe and record antitumor activity.

CORRELATIVE OBJECTIVES:

I. To evaluate the changes in the tumor immune microenvironment (exhausted T-cell phenotypes, percent T regulatory cells [T regs], T-cell activation) in peripheral blood and bone marrow caused by the addition of iberdomide to teclistamab and how they relate to minimal residual disease (MRD) status, responses rates and survival outcomes.

II. To evaluate soluble B-cell maturation antigen (sBCMA) levels at baseline and how they correlate to response rates and survival outcomes in patients treated with teclistamab plus iberdomide.

III. To identify the immunophenotypic and transcriptomic characterization of malignant plasma cells that are resistant to teclistamab and iberdomide.

OUTLINE: This is a dose-escalation study of iberdomide in combination with teclistamab.

Patients receive teclistamab subcutaneously (SC) on days 1, 4, 7, 15 and 22 for cycle 1 and days 1, 8, 15 and 22 for subsequent cycles. Patients also receive iberdomide orally (PO) once daily (QD) on days 1-21 for cycle 2 and beyond. Cycles repeat every 28 days for up to 4 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood and urine sample collection, bone marrow aspiration and biopsy and positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MR) throughout the trial.

After completion of study treatment, patients are followed up every 3-6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed multiple myeloma (MM), as defined in the International Myeloma Working Group (IMWG) criteria
* If patients have undergone autologous stem cell transplant (SCT), day 0 of SCT must be > 100 days to be eligible for the study
* Patients must have had disease progression after ≥ 4 prior lines of anti-myeloma treatments including one proteasome inhibitor (e.g., bortezomib, carfilzomib, ixazomib), one immunomodulatory imide drug (ImiD) (e.g., thalidomide, lenalidomide, pomalidomide [POM]), and one anti-CD38 monoclonal antibody (e.g., daratumumab, isatuximab)
* Patients must have measurable disease, defined as:

  * Serum M-protein ≥ 0.5 g/dL (≥ 5 g/L)
  * Urine M-protein ≥ 200 mg/24 h
  * Serum free light chain (FLC) assay: "involved" FLC level ≥ 10 mg/dL (≥ 100 mg/L) and an abnormal serum free light chain ratio (< 0.26 or > 1.65)
  * Note: Patients with non-secretory disease will be allowed to participate
* Age ≥ 18 years

  * Because no dosing or adverse event data are currently available on the use of iberdomide in combination with teclistamab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60)
* Hemoglobin ≥ 7.0 g/dL (≤ 28 days prior to registration) (Without growth factor support, blood transfusion, or platelet stimulating agents for the past 7 days, excluding erythropoietin)
* Absolute neutrophil count ≥ 1,000/mcL (≤ 28 days prior to registration) (Without growth factor support, blood transfusion, or platelet stimulating agents for the past 7 days, excluding erythropoietin)
* Platelets ≥ 50,000/mcL (≤ 28 days prior to registration) (Without growth factor support, blood transfusion, or platelet stimulating agents for the past 7 days, excluding erythropoietin)
* Total bilirubin ≤ 2 x institutional upper limit of normal (ULN) (≤ 28 days prior to registration)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN (≤ 28 days prior to registration)
* Estimated glomerular filtration rate (eGFR) > 30 mL/min (≤ 28 days prior to registration)
* Spot urine (albumin/creatine ratio) ≤ 500mg/g (56 mg/mmol) OR urine dipstick negative/trace (if > 1+ only eligible if confirmed ≤ 500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void) (≤ 28 days prior to registration)
* Note: Laboratory results obtained during screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the investigator may re-test the subject and the subsequent within range screening result may be used to confirm eligibility
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging done a minimum of 28 days after completion of central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Based on the mechanism of action, teclistamab may cause fetal harm when administered to a pregnant woman. Females of child-bearing potential (FCBP): should use effective contraception during treatment with teclistamab and for 5 months after the last dose. FCBP should not breast feed during treatment with teclistamab and for 5 months after the last dose. Should a FCBP become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. The effects of iberdomide on the developing human fetus are unknown. However, IMiDs are known to be teratogenic. FCBP must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to starting iberdomide, and again within 24 hours. FCBP must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control-one highly effective method and one additional effective method-at the same time, at least 28 days before starting iberdomide, while taking iberdomide, and for 28 days following discontinuation from the study. Examples of highly effective methods are intrauterine device, hormonal contraceptives, tubal ligation, or partner's vasectomy. Examples of barrier method are male condom, diaphragm, or cervical cap. FCBP must also agree to ongoing pregnancy testing. Men must practice complete abstinence or agree to use a condom during sexual contact with FCBP while participating in the study, during dose interruptions, and for at least 28 days following discontinuation from the study, even if he has undergone a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risk of fetal exposure
* Men must agree to abstain from donating and semen or sperm while taking iberdomide, during dose interruptions, and for at least 28 days after the last dose of iberdomide. FCBP must agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period
* All patients must agree to abstain from donating blood products while taking iberdomide and for at least 28 days after the last dose of iberdomide
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study subjects
* Willingness to adhere to the study visit schedule and other protocol requirements and provide mandatory blood and bone marrow specimens for correlative research
* Willingness to return to the enrolling institution for follow-up

Exclusion Criteria:

* Patients who have active plasma cell leukemia, active amyloid light chain (AL) (primary) amyloidosis, active polyneurophathy, organomegaly, endocrinopathy, monoclonal gammopathy and skin changes (POEMS) syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, myeloma protein, and skin changes), and Waldenstrom macroglobulinemia are ineligible
* If a patient develops recurrent/refractory (R/R) disease while receiving the most recent line of therapy, there is no need for a washout period
* Patients who have had prior anti-BCMA directed bispecific antibody (BsAb) therapy exposure (prior treatment with anti-BCMA directed antibody drug conjugate, anti-BCMA-directed chimeric antigen receptor (CAR) T cell therapy, and prior non-BCMA-targeting BsAb are permitted)
* Patients who have had prior treatment with a cereblon E3 ligase modulator, including mezigdomide, iberdomide, and CFT7455 (all currently in clinical development)
* Patients who received plasmapheresis ≤ 7 days prior to registration
* Patients who received a prior allogeneic stem cell transplant. Autologous SCT is allowed
* Patients who received a live or live-attenuated vaccine ≤ 30 days prior to registration. Patients are allowed to receive a COVID-19 vaccine at any timepoint during protocol treatment
* Systemic active infection requiring treatment
* Any unresolved toxicity ≥ grade 2 from previous treatment except for alopecia or peripheral neuropathy up to grade 2
* Patients who have had any major surgery ≤ 4 weeks prior to registration
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make this protocol unreasonably hazardous
* Patients with evidence of active mucosal or internal bleeding
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if participant otherwise meets entry criteria
* Patients with known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to teclistamab or iberdomide, or any of the components of the study treatment
* Patients who are taking any anticancer therapy other than hormonal therapy (for prostrate or breast cancer) and palliative radiotherapy (defined as radiation to ≤ 3 sites of active multiple myeloma)
* Patients who require immunosuppressive medications including, but not limited to, systemic corticosteroids at doses exceeding 10 mg/day of prednisone or equivalent. Use of immunosuppressive medications for the management of iberdomide-related adverse events (AEs) or in subjects with contrast allergies is acceptable. In addition, use of inhaled, topical, intranasal corticosteroids or local steroid injection (e.g., intra-articular injection) is permitted. Temporary use of corticosteroids for concurrent illnesses (e.g., food allergies, computed tomography [CT] scan contrast hypersensitivity, pneumonia, etc.) are acceptable
* Patients who require medications that are strong inhibitors or inducers of CYP3A4/5
* Patients who are receiving any other investigational agents
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because iberdomide is a thalidomide analog and thalidomide is a known human teratogen. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with iberdomide, breastfeeding should be discontinued if the mother is treated with iberdomide. These potential risks may also apply to other agents used in this study
* Patients who are unable or unwilling to undergo protocol required thromboembolism prophylaxis are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) of iberdomide when combined with teclistamab | At 28 days
  The RP2D will be defined as the pharmacologically optimal dose of iberdomide that can be combined with teclistamab and will be selected based on all available pharmacokinetic, pharmacodynamic, target engagement, efficacy, safety and tolerability data.
Maximum tolerated dose (MTD) of iberdomide when combined with teclistamab | At 28 days
  The MTD will be is defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 8 new patients).

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 4 weeks after last dose of study treatment
  AEs will be described and graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns. The relationship of the AEs to the study treatment will be taken into consideration.
Overall response rate (ORR) | Up to 2 years after last dose of study treatment
  The ORR will be estimated by the total number of patients who achieve a stringent complete response, complete response, very good partial response, or partial response divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Minimal residual disease (MRD) negativity | Up to 2 years after last dose of study treatment
  MRD negativity will be summarized descriptively at each specified timepoint.
Progression-free survival (PFS) | From registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 2 years after last dose of study treatment
  The distribution of PFS will be estimated using the method of Kaplan-Meier.
Time to progression | From registration to the earliest date of documentation of disease progression, assessed up to 2 years after last dose of study treatment
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Duration of response (DOR) | From earliest documentation of disease response to disease progression, assessed up to 2 years after last dose of study treatment
  The distribution of DOR will be estimated using the method of Kaplan-Meier.
Overall survival (OS) | From registration to death due to any cause, assessed up to 2 years after last dose of study treatment
  The distribution of OS will be estimated using the method of Kaplan-Meier.

OTHER OUTCOMES:
Tumor immune microenvironment | Up to 2 years after last dose of study treatment
  Flow cytometry will be utilized to assess the tumor immune microenvironment in the bone marrow and peripheral blood at baseline and during active treatment at specified time points. Values over time will be summarized graphically and descriptively. Paired sample approaches (Wilcoxon signed rank test) will be used to assess differences over time. The relationship between changes over time in each measure with response outcome measures will be explored using Wilcoxon's rank sum test.
Soluble B-cell maturation antigen levels | At baseline
  Values over time will be summarized graphically and descriptively. Paired sample approaches (Wilcoxon signed rank test) for these types of quantitative measures will be used to assess differences over time. The relationship between changes over time in each measure with response outcome measures will be explored using Wilcoxon's rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo D Parrondo, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (13):
- United States (13):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm